CLINICAL TRIAL: NCT04859322
Title: The Effect of Lifestyle-induced Hepatic Steatosis on Glucagon-stimulated Amino Acid Turnover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malte Palm Suppli, MD (Other)
Collaborators: Section of Molecular Physiology, Department of Nutrition, Exercise and Sports, Faculty of Science, University of Copenhagen, Denmark (Unknown); Rigshospitalet, Denmark (Other); Department of Biomedical Sciences & NNF Center for Protein Research, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen, Denmark (Unknown); Novo Nordisk Foundation Center for Basic Metabolic Research, Faculty of Health, and Medical Sciences, University of Copenhagen, Copenhagen, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Malte Palm Suppli, MD, MD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SIRG-2
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Glucagon Resistance
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Glucagon; Insulin; Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Participants (Experimental): 20 healthy participants included in the arm for 3 experimental days each. On each experimental day infusions of stable isotope glucose (0,6 micromol/kg/min), glucagon (1 hour low; 0,6 ng/kg/min, 2 hours high; 4,0 ng/kg/min), somatostatin (450 micrograms/hour) and insulin (0,1 mU/kg/min) will be administered. Between the first two experimental days the participants will follow a sedentary lifestyle combined with a high-calorie diet intervention
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Glucagon — Pancreatic clamp
  Other Names: Insulin; Somatostatin; 6,6 H2-glucose

SUMMARY:
Many patients with type 2 diabetes exhibit elevated plasma concentrations of the glucose-mobilising pancreatic hormone glucagon; i.e. hyperglucagonaemia. This contributes to the hyperglycaemic state of the patients and is considered an important component in the pathophysiology of type 2 diabetes; but the mechanisms underlying this phenomenon remain unclear. The liver constitutes the main target organ of glucagon, and studies have shown that hyperglucagonaemia goes hand in hand with hyperaminoacidaemia and that both are associated with non-alcoholic fatty liver disease (NAFLD), independently of the presence of type 2 diabetes. In line with this, several recent studies support the existence of a feedback-cycle between the liver and the pancreatic alpha cells, governed by circulating glucagon and amino acids. The investigators hypothesise that the presence of hepatic steatosis results in hepatic glucagon resistance at the level of amino acid turnover, i.e. impaired glucagon-induced suppression of circulating amino acid concentrations. If this hypothesis proves correct, it would establish build-up of fat in the liver as a core mechanism underlying hyperglucagonaemia and, since the hyperglucagonemia is at least partly responsible for the fasting hyperglycaemia, as an important contributor to the hyperglycaemia of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Normal fasting plasma glucose and glycated haemoglobin (HbA1c) <42 mmol/mol
* Body mass index (BMI) between 18.5 and 25 kg/m2
* Haemoglobin >8.3 mmol/l
* Habitual diet in accordance with the Nordic Nutrition Recommendations
* Age between 20 and 65 years
* Oral and written informed consent

Exclusion Criteria:

* Diabetes
* First-degree relatives with diabetes
* Fasting plasma triacylglycerol indicating dyslipidemia (≥2 mmol/l)
* Nephropathy (estimated glomerular filtration rate (eGFR) <60 ml/min and/or microalbuminuria with an albumin to creatinine ratio of 30-300 μg/mg)
* Known liver disease and/or alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 × normal values
* Signs of liver fibrosis and/or steatosis evaluated by FibroScan (CAP value >2380 dB/m and/or kPa >65.0) and/or FIB-4 score (>1.45)
* >5% steatosis evaluated by MRI carried out before experimental Day A (see Methods)
* Use of medication
* Use of dietary protein supplementation or any other dietary supplements that cannot be paused during participation
* Excessive training habits, defined as >2 weekly strength and/or aerobic training sessions
* Pregnancy and/or breastfeeding
* Implanted metal objects incompatible with magnetic resonance imaging (MRI)
* Any condition that the investigator feels would interfere with trial completion

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Nadir of the total amino acid concentration during a two-hour high physiological glucagon infusion during a pancreatic clamp with somatostatin | depending on the nadir between time 60 minutes and time 180 minutes
  micromol/liter

SECONDARY OUTCOMES:
average slope of the curve describing the change in the total amino acid concentration during 'supraphysiological' glucagon infusion | between time 60 minutes and time 180 minutes
  micromol/liter/minute
the incremental area under the curve (iAUC) for total amino acid concentrations during 'supraphysiological' glucagon infusion | between time 60 minutes and time 180 minutes
  micromol/liter
the percentage change in amino acid concentration during the last hour of the 'supraphysiological' glucagon infusion as assessed by baseline subtracted AUC | between time 60 minutes and time 180 minutes
  micromol/liter

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Copenhagen, Denmark